CLINICAL TRIAL: NCT07213401
Title: Non-invasive Monitoring of Newborns in the First Hours of Life for the Prevention of SUPC (Sudden Unexpected Postnatal Collapse): Interventional Study With Medical Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, PI, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DARE_NEO_SUPC
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Sudden Unexpected Postnatal Collapse -SUPC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- newborn (Other): The study population will consist of all babies born in the delivery room with a gestational age of ³35 weeks who are considered suitable for SSC in the first 2 hours of life and subsequently for rooming-in according to clinical practice.
  Interventions: Device: ComfTech HOWDY BABY

INTERVENTIONS:
Device: ComfTech HOWDY BABY — The Comftech HOWDYBABY medical device is a device for monitoring vital physiological parameters, in particular for monitoring heart rate and respiratory rate, consisting of a sensor-equipped belt. Blood oxygen saturation can also be monitored using a compatible accessory.

SUMMARY:
The application of non-invasive monitoring via a wearable device in newborns during the first 48-72 hours of life could enable early recognition and timely management of episodes that may result in SUPC, thereby improving clinical practice.

DETAILED DESCRIPTION:
SUPC is a rare event, with maximum incidence in the first 2 hours of life of the newborn. Despite the rarity of events, the consequences can be dramatic, with a high risk of death and severe neurological disabilities. To date, prevention of events is based on serial clinical monitoring of newborns during skin-to-skin contact.

Some non-invasive monitoring systems integrated into wearable textiles have proven to be reliable and are well tolerated by newborns, families, and healthcare personnel.

The application of non-invasive monitoring via a wearable device in newborns during the first 48-72 hours of life could enable early recognition and timely management of episodes that may result in SUPC, thereby improving clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ³ 35 weeks
* Apgar score at 5 minutes ³ 8
* Acquisition of written informed consent from the parent/guardian

Exclusion Criteria:

* Major congenital malformations
* Family history of silver allergy

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
prodromal events of SUPC | 72 hours
  Measure how many prodromal events of SUPC (bradycardia, bradypnea, apnea) are detected with the ComfTech HOWDY BABY device (ComfTech S.r.l.), outside the times scheduled for clinical monitoring in the first 72 hours of life of newborns.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Aoubo, Bologna, BO, Italy